CLINICAL TRIAL: NCT07206992
Title: Assessment of a 24-hour Preoperative Course of Antibiotic Therapy for Endoscopic Urological Surgery in Case of Positive Urine Culture
Acronym: ANTIBIURO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-A01224-41
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Urologic Surgery
Keywords: Urologic Surgery Preoperative Antibiotic Therapy
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotic therapy 24 hours (Experimental): Antibiotic therapy will start 24 hours before urological surgery
  Interventions: Drug: 24 hours antibiotics
- Antibiotic therapy 48 hours (Active Comparator): Antibiotic therapy will start 48 hours before urological surgery
  Interventions: Drug: 48 hours antibiotics

INTERVENTIONS:
Drug: 24 hours antibiotics — Antibiotic therapy will start 24 hours before urological surgery
  Arms: Antibiotic therapy 24 hours
Drug: 48 hours antibiotics — Antibiotic therapy will start 48 hours before urological surgery
  Arms: Antibiotic therapy 48 hours

SUMMARY:
Endourology poses the problem of post-operative infections. The need to obtain a negative urine culture prior to surgery is accepted, and the effectiveness of this measure in reducing the risk of post-operative infection has been proven.

Current French recommendations are unanimous in favour of preventive treatment for asymptomatic bacteriuria (positive urine culture) prior to urological procedures involving contact with urine. These same recommendations specify that treatment should be brief, with a preoperative course of antibiotics lasting 48 hours.

However, the scientific literature on the subject does not provide an answer to the question of whether 48 hours is the optimal duration of preoperative antibiotic treatment to avoid the risk of postoperative infection.

In this context, it is interesting to evaluate a duration of preoperative antibiotic therapy limited to 24 hours, as no study can confirm that 24 hours of treatment is insufficient to prevent post-operative infection.

DETAILED DESCRIPTION:
Endourology poses the problem of post-operative infections. The need to obtain a negative urine culture prior to surgery is accepted, and the effectiveness of this measure in reducing the risk of post-operative infection has been proven.

Current French recommendations are unanimous in favour of preventive treatment for asymptomatic bacteriuria (positive urine culture) prior to urological procedures involving contact with urine. These same recommendations specify that treatment should be brief, with a preoperative course of antibiotics lasting 48 hours.

However, the scientific literature on the subject does not provide an answer to the question of whether 48 hours is the optimal duration of preoperative antibiotic treatment to avoid the risk of postoperative infection. Studies have shown that a single parenteral administration of antibiotics in the context of asymptomatic bacteriuria prior to urological surgery is effective in preventing post-operative infection. Furthermore, in some practical situations related to the time taken for the laboratory to return urine culture results, preoperative antibiotic therapy has been limited to 24 hours without any infections developing.

In this context, it is interesting to evaluate a duration of preoperative antibiotic therapy limited to 24 hours, as no study can confirm that 24 hours of treatment is insufficient to prevent post-operative infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients scheduled for urological endoscopy for one of the following indications: endoscopic surgery of the upper urinary tract (diagnostic, for treatment of stones or ureteral strictures), endoscopic prostate surgery (with or without laser: enucleation, vaporisation, resection), endoscopic surgery of the bladder and urethra (particularly tumours, strictures and foreign bodies) and ureteral stent surgery
* Patients with a positive preoperative urine culture (presence of bacteria at more than 103/mL)
* Asymptomatic patients (no signs of urinary tract infection in particular)
* Patients affiliated with or covered by a social security scheme
* French-speaking patients who have signed an informed consent form

Exclusion Criteria:

* Patient participating in another clinical trial
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Patient with an immune deficiency
* Patient presenting symptoms of preoperative pyelonephritis (fever)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 894 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative infectious complications. | One month
  Post-operative infectious complications will be assessed as %. Post-operative infection will be defined as:
  • A fever (T>38°C) / hypothermia (T<36°C) with no other cause other than urological, OR lower back pain, OR lower urinary tract symptoms that appeared or persisted at least 7 days after the procedure.
  AND
  • A positive urine culture (leukocyturia >or= 10^4/ml and positive urine culture >10^3 cfu/ml for a uropathogen)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé des Peupliers, Paris, France

IPD SHARING:
Plan to Share IPD: No